CLINICAL TRIAL: NCT04337307
Title: Evaluation of Two Procedures of Incubator's Decontamination in a NICU
Brief Title: Decontamination of Incubators in a NICU (Neonatal Intensive Care Unit)
Acronym: DECONTA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0299; ID-RCB (Other: 2020-A00818-31)
Record Dates: First submitted 2020-04-02; First posted 2020-04-07 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Health Care Worker Patient Transmission
Keywords: Bacterial colonization of incubators

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard decontamination: incubators decontaminated with antiseptic molecules, healthcare workers involved in this decontamination, patients housed in these incubators
  Interventions: Biological: Skin sampling of the hands of the healthcare workers involved in the decontamination of incubators
- steam pulverization: incubators decontaminated with steam pulverization, healthcare workers involved in this decontamination, patients housed in these incubators
  Interventions: Biological: Skin sampling of the hands of the healthcare workers involved in the decontamination of incubators

INTERVENTIONS:
Biological: Skin sampling of the hands of the healthcare workers involved in the decontamination of incubators — Each incubator will be sampled in 5 points before and after decontamination. The healthcare worker that will be involved in the decontamination will also be sampled (skin sample of the hand) before and after decontamination of the incubator.
  All the samples will be analyzed for the presence of pathogenic bacteria, using an inoculation on selective agar then an identification of each bacterial colony.

SUMMARY:
Nosocomial infections are responsible for morbidity and mortality in hospitalized neonates. The environment of the neonates and especially the incubators can constitute the reservoir of pathogenic bacteria. That is why decontamination of incubators is a major step in the fight against nosocomial infections in NICUs.

The hypothesize is that the usual procedure of decontamination, based on antiseptic molecules, is not sufficient to eradicate all pathogenic bacteria from the incubators.

In this study the investigator's aim to assess the efficacy of the usual procedure of decontamination and to compare it with another procedure based on steam pulverization. Another objective will be to explore a possible contamination of the hands of the healthcare workers, that can be involved in the cycle of transmission of bacteria to neonates. Finally, clinical data about the neonates housed in the incubator will be retrieved from clinical reports, to identify the occurrence of sepsis and if so, to compare the bacteria involved in the sepsis and the bacteria present in the incubator.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers involved in the decontamination process of incubators during the study period (period of sampling of incubators before and after decontamination)
* The two people involved in the sampling of incubators
* The patients (neonates) that will be housed in one incubator decontaminated and sampled during the study period

Exclusion Criteria:

* Refusal to participate for healthcare workers and people involved in the sampling
* Refusal to give access to the clinical data of his child for the parent of the patients included in the study-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare workers of the NICU of the Hopital Femme Mere enfant (HFME), Hospices Civils de Lyon, that will be involved in the process of decontamination of the incubators during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Absence of bacterial contamination | Day 0 (just before the decontamination)
  Efficacy of decontamination will be defined for each incubator as the absence of bacterial contamination after the process of decontamination
Absence of bacterial contamination | Day 0 (just after the decontamination)
  Efficacy of decontamination will be defined for each incubator as the absence of bacterial contamination after the process of decontamination

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France